CLINICAL TRIAL: NCT04608747
Title: Effect of Tahini Consumption on Oxidative Stress and Inflammation Markers as Well as Endothelial Function and Arterial Stiffness in Healthy Volunteers
Brief Title: Tahini, Antioxidant Status and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, PANAGIOTIS KANELLOS, POSTDOCTORAL RESEARCHER, Harokopio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 703
Record Dates: First submitted 2020-10-25; First posted 2020-10-29 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Oxidative Stress; Endothelial Function; Blood Pressure; Arterial Stiffness; Blood Glucose
Keywords: tahini; sesame; antioxidants; postprandial
MeSH Terms: conditions — SeSAME syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): After an overnight fast, participants subjected to baseline measurements and blood and urine collection and then consumed an amount of 50 g of tahini. Blood and urine collection and other measurements were repeated 4 h postprandially.
  Interventions: Other: Tahini

INTERVENTIONS:
Other: Tahini — Fifty grams of tahini were consumed by 20 healthy males

SUMMARY:
Cardiovascular disease (CVD), a cluster of disorders that affect heart and blood vessels, is the leading cause of morbidity and mortality around the world and is responsible for 17.9 million deaths annually worldwide. CVD risk factors can be modifiable (nutrition, physical activity, obesity, smoking, hyperlipidemia, hypertension and diabetes) and non-modifiable (age, gender, ethnicity, family history and socioeconomic status). Chronic exposure to CVD risk factors induces oxidative stress and promotes inflammation. In addition, endothelial cells in response to the inflammatory reaction secrete growth factors, leading to the destruction of vascular endothelium and promoting atherogenesis.

Oxidative stress refers to the imbalance between anti-oxidant and pro-oxidant compounds, with predominance of the pro-oxidant ones. Reactive Oxygen Species overproduction has been implicated in pathogenesis and complications of numerous diseases including diabetes, cardiovascular diseases, cancer, neurodegenerative diseases and chronic kidney disease.

Moreover, endothelium consists of a single layer of endothelial cells; it is the natural barrier between blood and tissues and also an endocrine organ. It plays a key role in vascular homeostasis by maintaining a balance between vasodilation and vasoconstriction and is responsible for fluid filtration, blood vessel tone, hormone trafficking, hemostasis, regulation of blood flow and growth of blood vessels. Thus, reductions in endothelial function are detrimental and predict and precede the development of overt CVD.

Sesame belongs to Pedaliaceae family and can be consumed in different forms such as seeds, oil or tahini, i.e., a 100 % peeled, ground and roasted sesame paste. Sesame seeds are rich in polyunsaturated fatty acids, proteins, vitamin E and lignans, such as sesamin, sesamolin and sesamol. Recent studies have highlighted the antioxidant, antihypertensive, hypolipidemic and appetite control properties of sesame seeds and sesame oil.

Regarding the consumption of tahini and its effect on human health, only three studies are available in the current literature, one of them in patients with type 2 diabetes, one in diabetic animal model and one in Alzheimer's disease animal model. Thus, the aim of the present study is to investigate the effect of tahini consumption on oxidative stress, blood pressure, endothelial function and arterial stiffness in healthy males postprandially.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD), a cluster of disorders that affect heart and blood vessels, is the leading cause of morbidity and mortality around the world and is responsible for 17.9 million deaths annually worldwide. CVD includes coronary heart disease, peripheral arterial disease, cerebrovascular disease, rheumatic heart disease, congenital heart disease, deep vein thrombosis and pulmonary embolism. CVD risk factors can be modifiable (nutrition, physical activity, obesity, smoking, hyperlipidemia, hypertension and diabetes) and non-modifiable (age, gender, ethnicity, family history and socioeconomic status). Chronic exposure to CVD risk factors induces oxidative stress and promotes inflammation. In addition, endothelial cells in response to the inflammatory reaction secrete growth factors, leading to the destruction of vascular endothelium and promoting atherogenesis.

Oxidative stress refers to the imbalance between anti-oxidant and pro-oxidant compounds, with predominance of the pro-oxidant ones. These compounds are also called Reactive Oxygen Species (ROS) or free radicals and are unstable atoms or molecules. Their generation, as products of normal cellular metabolism, occurs naturally by endogenous sources (e.g. mitochondria, peroxisomes and endoplasmic reticulum) through enzymatic and non-enzymatic reactions. Furthermore, exogenous sources implicated in free radical production are air pollution, alcohol consumption, tobacco smoking, ultraviolet light exposure, industrial solvents and others. Free radical production is regulated by the well-organized human endogenous enzymatic and non-enzymatic antioxidant system, along with the exogenous antioxidants found in food. However, in some cases antioxidant system fails to eliminate ROS overproduction and can consequently induce serious damage to important for life biomolecules (DNA, lipids, proteins), leading to cell injury and death. Thus, ROS overproduction has been implicated in pathogenesis and complications of numerous diseases including diabetes, cardiovascular diseases, cancer, neurodegenerative diseases and chronic kidney disease.

Moreover, endothelium consists of a single layer of endothelial cells; it is the natural barrier between blood and tissues and also an endocrine organ. It plays a key role in vascular homeostasis by maintaining a balance between vasodilation and vasoconstriction. Moreover, vascular endothelium is responsible for fluid filtration, blood vessel tone, hormone trafficking, hemostasis, regulation of blood flow and growth of blood vessels. Thus, reductions in endothelial function are detrimental and predict and precede the development of overt CVD.

Sesame belongs to Pedaliaceae family and can be consumed in different forms such as seeds, oil or tahini, i.e., a 100 % peeled, ground and roasted sesame paste. Sesame seeds are rich in polyunsaturated fatty acids (PUFAs), proteins, vitamin E and lignans, such as sesamin, sesamolin and sesamol. Recent studies have highlighted the antioxidant, antihypertensive, hypolipidemic and appetite control properties of sesame seeds and sesame oil. Moreover, few studies have investigated the effect of sesame consumption on blood pressure, endothelial function and arterial stiffness in human population. According to a metanalysis, sesame consumed in form of seed, oil, capsule or bar decreased both systolic blood pressure (SBP) and diastolic blood pressure (DBP), while sesame oil consumption was found to improve endothelial function both in the postprandial state and after long term consumption in hypertensive men.

Regarding the consumption of tahini and its effect on human health, only three studies are available in the current literature, one of them in patients with type 2 diabetes, one in diabetic animal model and one in Alzheimer's disease animal model. Thus, the aim of the present study is to investigate the effect of tahini consumption on oxidative stress, blood pressure, endothelial function and arterial stiffness in healthy males postprandially.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 40 years
* Body Mass Index (BMI)<30 kg/m2

Exclusion Criteria:

* alcohol or drug abuse,
* any medication or vitamin/mineral supplementation
* alternative diet (vegetarian, macrobiotic, etc.)
* recent use of antibiotics
* history of any chronic disease

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Concentration of oxidative stress biomarkers | Four hours after tahini consumption
  concentration of urinary 8-iso-prostaglandin F2a

CONTACTS AND LOCATIONS:
Overall Officials: NIKOLAOS K TENTOLOURIS, PROF, Study Director — Diabetes CeMedical School, National and Kapodistrian University of Athens, Laiko General Hospital
Locations (1):
- Diabetes Center, First Department of Propaedeutic Internal Medicine, Medical School, National and Kapodistrian University of Athens, Laiko General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sies H. Oxidative stress: a concept in redox biology and medicine. Redox Biol. 2015;4:180-3. doi: 10.1016/j.redox.2015.01.002. Epub 2015 Jan 3. PMID 25588755
- [Background] Kumar, S., & Pandey, A. (2015). Free Radicals: Health Implications and their Mitigation by Herbals. British Journal Of Medicine And Medical Research, 7(6), 438-457. doi: 10.9734/bjmmr/2015/16284
- [Background] Phaniendra A, Jestadi DB, Periyasamy L. Free radicals: properties, sources, targets, and their implication in various diseases. Indian J Clin Biochem. 2015 Jan;30(1):11-26. doi: 10.1007/s12291-014-0446-0. Epub 2014 Jul 15. PMID 25646037
- [Background] Birben E, Sahiner UM, Sackesen C, Erzurum S, Kalayci O. Oxidative stress and antioxidant defense. World Allergy Organ J. 2012 Jan;5(1):9-19. doi: 10.1097/WOX.0b013e3182439613. Epub 2012 Jan 13. PMID 23268465
- [Background] Willcox JK, Ash SL, Catignani GL. Antioxidants and prevention of chronic disease. Crit Rev Food Sci Nutr. 2004;44(4):275-95. doi: 10.1080/10408690490468489. PMID 15462130
- [Background] Ravarotto V, Simioni F, Pagnin E, Davis PA, Calo LA. Oxidative stress - chronic kidney disease - cardiovascular disease: A vicious circle. Life Sci. 2018 Oct 1;210:125-131. doi: 10.1016/j.lfs.2018.08.067. Epub 2018 Aug 31. PMID 30172705
- [Background] Zoumpoulakis, P., Sinanoglou, V., Batrinou, A., Strati, I., Miniadis-Meimaroglou, S., & Sflomos, K. (2012). A combined methodology to detect γ-irradiated white sesame seeds and evaluate the effects on fat content, physicochemical properties and protein allergenicity. Food Chemistry, 131(2), 713-721. doi: 10.1016/j.foodchem.2011.09.049
- [Background] Namiki M. Nutraceutical functions of sesame: a review. Crit Rev Food Sci Nutr. 2007;47(7):651-73. doi: 10.1080/10408390600919114. PMID 17943496
- [Background] Raeisi-Dehkordi, H., Mohammadi, M., Moghtaderi, F., & Salehi-Abargouei, A. (2018). Do sesame seed and its products affect body weight and composition? A systematic review and meta-analysis of controlled clinical trials. Journal Of Functional Foods, 49, 324-332. doi: 10.1016/j.jff.2018.08.036
- [Background] Pathak N, Rai AK, Kumari R, Bhat KV. Value addition in sesame: A perspective on bioactive components for enhancing utility and profitability. Pharmacogn Rev. 2014 Jul;8(16):147-55. doi: 10.4103/0973-7847.134249. PMID 25125886
- [Background] Gouveia Lde A, Cardoso CA, de Oliveira GM, Rosa G, Moreira AS. Effects of the Intake of Sesame Seeds (Sesamum indicum L.) and Derivatives on Oxidative Stress: A Systematic Review. J Med Food. 2016 Apr;19(4):337-45. doi: 10.1089/jmf.2015.0075. PMID 27074618
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Park KH, Park WJ. Endothelial Dysfunction: Clinical Implications in Cardiovascular Disease and Therapeutic Approaches. J Korean Med Sci. 2015 Sep;30(9):1213-25. doi: 10.3346/jkms.2015.30.9.1213. Epub 2015 Aug 13. PMID 26339159
- [Background] Kruger-Genge A, Blocki A, Franke RP, Jung F. Vascular Endothelial Cell Biology: An Update. Int J Mol Sci. 2019 Sep 7;20(18):4411. doi: 10.3390/ijms20184411. PMID 31500313
- [Background] Rajendran P, Rengarajan T, Thangavel J, Nishigaki Y, Sakthisekaran D, Sethi G, Nishigaki I. The vascular endothelium and human diseases. Int J Biol Sci. 2013 Nov 9;9(10):1057-69. doi: 10.7150/ijbs.7502. eCollection 2013. PMID 24250251
- [Background] Alipoor B, Haghighian MK, Sadat BE, Asghari M. Effect of sesame seed on lipid profile and redox status in hyperlipidemic patients. Int J Food Sci Nutr. 2012 Sep;63(6):674-8. doi: 10.3109/09637486.2011.652077. Epub 2012 Jan 23. PMID 22263599
- [Background] Khosravi-Boroujeni H, Nikbakht E, Natanelov E, Khalesi S. Can sesame consumption improve blood pressure? A systematic review and meta-analysis of controlled trials. J Sci Food Agric. 2017 Aug;97(10):3087-3094. doi: 10.1002/jsfa.8361. Epub 2017 May 12. PMID 28387047
- [Background] Kamal-Eldin A, Frank J, Razdan A, Tengblad S, Basu S, Vessby B. Effects of dietary phenolic compounds on tocopherol, cholesterol, and fatty acids in rats. Lipids. 2000 Apr;35(4):427-35. doi: 10.1007/s11745-000-541-y. PMID 10858028
- [Background] Wu WH, Kang YP, Wang NH, Jou HJ, Wang TA. Sesame ingestion affects sex hormones, antioxidant status, and blood lipids in postmenopausal women. J Nutr. 2006 May;136(5):1270-5. doi: 10.1093/jn/136.5.1270. PMID 16614415
- [Background] Khalesi S, Paukste E, Nikbakht E, Khosravi-Boroujeni H. Sesame fractions and lipid profiles: a systematic review and meta-analysis of controlled trials. Br J Nutr. 2016 Mar 14;115(5):764-73. doi: 10.1017/S0007114515005012. Epub 2016 Jan 13. PMID 26758593
- [Background] Hirata F, Fujita K, Ishikura Y, Hosoda K, Ishikawa T, Nakamura H. Hypocholesterolemic effect of sesame lignan in humans. Atherosclerosis. 1996 Apr 26;122(1):135-36. doi: 10.1016/0021-9150(95)05769-2. No abstract available. PMID 8724120
- [Background] Neves Ribeiro D, Goncalves Alfenas Rde C, Bressan J, Brunoro Costa NM. The effect of oilseed consumption on appetite and on the risk of developing type 2 diabetes mellitus. Nutr Hosp. 2013 Mar-Apr;28(2):296-305. doi: 10.3305/nh.2013.28.2.6309. PMID 23822678
- [Background] Karatzi K, Stamatelopoulos K, Lykka M, Mantzouratou P, Skalidi S, Zakopoulos N, Papamichael C, Sidossis LS. Sesame oil consumption exerts a beneficial effect on endothelial function in hypertensive men. Eur J Prev Cardiol. 2013 Apr;20(2):202-8. doi: 10.1177/2047487312437625. Epub 2012 Jan 25. PMID 22345690